CLINICAL TRIAL: NCT05401474
Title: Assessing Recruitability for Flow Individualization in Patients Treated With Nasal High Flow: a Physiological Study (The iFLOW Study)
Brief Title: Individualization Flow in Patients Treated With High Flow Nasal Therapy (iFLOW)
Acronym: iFLOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PR(AG)21/2022
Record Dates: First submitted 2022-04-05; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: High-Flow Nasal Cannula; Oxygen Therapy; Acute Respiratory Failure; Respiratory Failure; Lung Injury
Keywords: High-Flow Nasal Cannula; Oxygen therapy; Electrical Impedance Tomography; Lung injury; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency; Lung Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30 L/min (Active Comparator): HFNC at 30L/min. FiO2 adjusted to reach SpO2 95%
  Interventions: Device: High Flow Nasal Cannula at 30L/min
- 45 L/min (Experimental): HFNC at 45L/min. FiO2 adjusted to reach SpO2 95%
  Interventions: Device: High Flow Nasal Cannula at 45L/min
- 60 L/min (Experimental): HFNC at 60L/min. FiO2 adjusted to reach SpO2 95%
  Interventions: Device: High Flow Nasal Cannula at 60L/min

INTERVENTIONS:
Device: High Flow Nasal Cannula at 30L/min — Flow will be set at 30L/min, FiO2 will be adjusted manually to maintain SpO2within the target range
  Arms: 30 L/min
Device: High Flow Nasal Cannula at 45L/min — Flow will be set at 45L/min, FiO2 will be adjusted manually to maintain SpO2within the target range
  Arms: 45 L/min
Device: High Flow Nasal Cannula at 60L/min — Flow will be set at 60L/min, FiO2 will be adjusted manually to maintain SpO2within the target range
  Arms: 60 L/min

SUMMARY:
In patients with acute hypoxemic respiratory failure (AHRF), High Flow Nasal Therapy (HFNT) improves oxygenation, tolerance, and decreases work of breathing as compared to standard oxygen therapy by facemask.

The hypothesis is that this flow challenge (ROX index variation from 30 to 60L/min) could be used as a test for assessing changes in lung aeration, analyzed by the variation in end expiratory lung volume (ΔEELV), in patients treated with HFNC. It may allow to personalize the flow settings during HFNC. In this sense, an increase in EELV will be observed with higher flows in responders and, therefore, these participants may benefit from increasing the flow. In contrast, to increase the flow in non-responders (no significant increase in EELV with higher flows) increase the risk of patient self-inflicted lung injury (P-SILI).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to the ICU requiring NHF due to AHRF that will be defined as an SpO2/FIO2 ratio <315

Exclusion Criteria:

* Patient with indication for immediate CPAP, NIV, or invasive mechanical ventilation
* Hemodynamic instability defined as a need of continuous infusion of epinephrine or norepinephrine > 1 mg/h
* Severe acidosis (pH ≤ 7.25)
* Pregnant woman
* Tracheotomised patient
* Formalized ethical decision to withhold or withdraw life support
* Patient under guardianship
* Patient deprived of liberties
* Patient already enrolled in the present study in a previous episode of acute respiratory failure
* Patient who does not consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-11-05 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
To validate the correlation between the change in ROX index and the change in EELV | 20 minutes
  Change in ROX is defined as the difference in ROX index (SpO2/FiO2/respiratory rate) between 2 flows. Change in EELV is the difference in End-Expiratory Lung Volume as determined by EIT.

SECONDARY OUTCOMES:
To assess the changes in aeration distribution (by the variable center of ventilation (CoV)) measured by EIT at different flows (30L/min, 45 L/min and 60L/min). | 20 minutes
  Lung aeration as defined by the variable center of ventilation (CoV) in EIT.
To assess the changes in lung homogeneity (by the variable global inhomogeneity index (GI)) measured by EIT at differents flows (30L/min, 45 L/min and 60L/min). | 20 minutes
  Lung homogeneity as defined by global inhomogeneity index (GI) by EIT
To analyze the differences in SpO2 at different flows | 20 minutes
  SpO2 by pulseoxymetry
To analyze the differences in respiratory rate at different flows | 20 minutes
  Breaths/minute
To analyze the differences in the FiO2 used at different flows | 20 minutes
  FiO2 will be titrated manually to achieve a predefined SpO2 range (92 - 96%; 88-92% for patients with chronic respiratory disease)
To analyze the differences in patient comfort at different flows, using the visual analogic scale (from 0 to 10) | 20 minutes.
  Comfort score by visual analogic scale. From 0 (worst outcome) to 10 (best outocome).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricard JD, Roca O, Lemiale V, Corley A, Braunlich J, Jones P, Kang BJ, Lellouche F, Nava S, Rittayamai N, Spoletini G, Jaber S, Hernandez G. Use of nasal high flow oxygen during acute respiratory failure. Intensive Care Med. 2020 Dec;46(12):2238-2247. doi: 10.1007/s00134-020-06228-7. Epub 2020 Sep 8. PMID 32901374
- [Background] Mauri T, Alban L, Turrini C, Cambiaghi B, Carlesso E, Taccone P, Bottino N, Lissoni A, Spadaro S, Volta CA, Gattinoni L, Pesenti A, Grasselli G. Optimum support by high-flow nasal cannula in acute hypoxemic respiratory failure: effects of increasing flow rates. Intensive Care Med. 2017 Oct;43(10):1453-1463. doi: 10.1007/s00134-017-4890-1. Epub 2017 Jul 31. PMID 28762180
- [Background] Roca O, Messika J, Caralt B, Garcia-de-Acilu M, Sztrymf B, Ricard JD, Masclans JR. Predicting success of high-flow nasal cannula in pneumonia patients with hypoxemic respiratory failure: The utility of the ROX index. J Crit Care. 2016 Oct;35:200-5. doi: 10.1016/j.jcrc.2016.05.022. Epub 2016 May 31. PMID 27481760
- [Background] Bachmann MC, Morais C, Bugedo G, Bruhn A, Morales A, Borges JB, Costa E, Retamal J. Electrical impedance tomography in acute respiratory distress syndrome. Crit Care. 2018 Oct 25;22(1):263. doi: 10.1186/s13054-018-2195-6. PMID 30360753